CLINICAL TRIAL: NCT01089920
Title: Dose Response Bioavailability of Coffee and Green Tea Antioxidants in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 09.06.MET
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Tea; Coffee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- High dose coffee (Experimental): High dose of polyphenols from soluble coffee
  Interventions: Other: Coffee
- Medium dose coffee (Experimental): Medium dose of polyphenols from soluble coffee
  Interventions: Other: Coffee
- Low dose coffee (Experimental): Low dose of polyphenols from soluble coffee
  Interventions: Other: Coffee
- High dose green tea (Experimental): High dose of green tea polyphenols from infusion
  Interventions: Other: Green tea
- Medium dose green tea infusion (Experimental): Medium dose of green polyphenols from infusion
  Interventions: Other: Green tea
- Low dose green tea infusion (Experimental): low dose of polyphenols from an infusion of green tea
  Interventions: Other: Green tea

INTERVENTIONS:
Other: Green tea — Infusion (tea bags) from commercially available green tea
  Arms: High dose green tea; Low dose green tea infusion; Medium dose green tea infusion
Other: Coffee — Soluble coffee commercially available
  Other Names: Soluble coffee
  Arms: High dose coffee; Low dose coffee; Medium dose coffee

SUMMARY:
Coffee and green tea are 2 widely consumed beverages. Both contain polyphenol antioxidant compounds (chlorogenic acids for coffee and catechins for tea). The bioavailability of catechins is somewhat known and has been referenced in the literature. However, bioavailability data from tea infusion is non-existent, even though it reflects better how consumers drink this beverage. In addition, bioavailability of coffee chlorogenic acids is less understood and no dose response study has been reported so far in the literature. Thus, there is a great need to understand and reinforce our knowledge on the bioavailability of coffee and tea polyphenol compounds.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years, male and female
* Healthy as determined by the medical questionnaire and the medical visit
* Normal weight: BMI 18 - 25
* Coffee drinkers with an average consumption of 2-5 cups per day
* Having given informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases / disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer
* Have had a gastrointestinal surgery, except appendicectomy
* Difficulty to swallow
* Have a regular consumption of medication
* Have taken antibiotic therapy within the last 6 months
* Alcohol consumption > 2 units a day
* Smokers (more than 5 cigarettes per day)
* Have given blood within the last 3 weeks
* Volunteers who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 3 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Compare plasma Area under the curve (AUC) of highest and lowest dose of coffee for chlorogenic and phenolic acid metabolites | Measurements done over 24h after ingestion

SECONDARY OUTCOMES:
Compare Area under the curve (AUC), Maximum plasma concentration (Cmax), Time to reach maximum plasma concentration (Tmax) and half-life (T1/2) of all three doses of coffee for chlorogenic and phenolic acid metabolites | Measurements done over 12h after ingestion
Compare AUC, Cmax, Tmax and T1/2 of all three doses of green tea for catechin metabolites | Measurements done over 12h after ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, M.D., Ph.D., Principal Investigator — Nestec
Locations (1):
- Nestle Research Center, Lausanne, Switzerland